CLINICAL TRIAL: NCT04034771
Title: The Effect of Melatonin Administration on Sedation Level as Adjuvant to Propofol in Mechanically Ventilated Traumatic Brain Injury Patient: RCT
Brief Title: The Effect of Melatonin Administration on Sedation Level as Adjuvant to Propofol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mahmoud salem soliman, dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: sedation in TBI
Record Dates: First submitted 2019-07-23; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: melatonin
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Melatonin; Tablets; Propofol

STUDY DESIGN:
Who Masked: Participant
Masking Description: patient will be under general sedation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol and melatonin (Experimental): propofol iv infusion and melatonin 10 mg tablet through a nasogastric tube, once at admission.
  Interventions: Drug: Melatonin 10 MG Oral Tablet; Drug: Propofol
- propofol and placebo (Active Comparator): propofol iv infusion and a placebo tablets through a nasogastric tube once at admission
  Interventions: Drug: Propofol; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Melatonin 10 MG Oral Tablet — Melatonin tablets
  Other Names: circadian
  Arms: propofol and melatonin
Drug: Propofol — propofol amp
  Other Names: diprivan
Drug: Placebo oral tablet — sugar pill manufactured to mimic melatonin tablets
  Other Names: palacebo tabletes (for melatonin)
  Arms: propofol and placebo

SUMMARY:
This study assess the effect of administration of exogenous melatonin as adjuvant to propofol on the level of sedation and consequently the rate of propofol infusion.

DETAILED DESCRIPTION:
38 patients with traumatic brain injuries requiring mechanical ventilation and sedation were randomly allocated to two groups (melatonin group)19 patients and (control group)19 patients. In both groups a bolus of propofol 1mglkg was given by titration till the patient reached a sedation level value of (60-70) on the bispectral index (BIS), Then propofol infusion started at a rate of 1mglkglhr as a maintenance and rate adjusted according to our targeted sedation level, melatonin 10 mg tablet was crushed and mixed with 20 ml of water and administrated through a nasogastric tube followed by another 20 ml to flush out the residue for (melatonin group). While (control Group) received a placebo tablets by the same wayBIS value and propofol infusion rate was recorded over 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age group from 18 to 65
* Both sexes
* Patients on a mechanical ventilation and need sedation
* Patients who are vitally stable

Exclusion Criteria:

* Gastro intestinal tract impractabililty
* Pregnant female
* Vitally unstable patients who cannot tolerate propofol infusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
level of sedation | 6 hours
  observe the effect of the oral administration of 10 mg melatonin on decreasing the dose of propofol infusion in a mechanically ventilated patient with a traumatic brain injury using bispectral index

SECONDARY OUTCOMES:
• Arterial blood pressure | 6 hours
  measuring Blood pressure in mmgh just before and after start of propofol infusion and every hour for successive 6 hours
Heart rate | Measuring the heart rate as beats per minutes just before and after propofol infusion and every hour for the next 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud s Soliman, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr Alini Univeristy Hospital, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP
Time Frame: one month
Access Criteria: open

REFERENCES:
- [Background] Samarkandi A, Naguib M, Riad W, Thalaj A, Alotibi W, Aldammas F, Albassam A. Melatonin vs. midazolam premedication in children: a double-blind, placebo-controlled study. Eur J Anaesthesiol. 2005 Mar;22(3):189-96. doi: 10.1017/s0265021505000335. PMID 15852991
- [Background] Yousaf F, Seet E, Venkatraghavan L, Abrishami A, Chung F. Efficacy and safety of melatonin as an anxiolytic and analgesic in the perioperative period: a qualitative systematic review of randomized trials. Anesthesiology. 2010 Oct;113(4):968-76. doi: 10.1097/ALN.0b013e3181e7d626. PMID 20823763